CLINICAL TRIAL: NCT00330733
Title: Salsalate Therapy to Reduce Insulin Resistance and Cardiovascular Risk
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLIN-011-05F
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Atherosclerosis; Cardiovascular Disease; Inflammation; Insulin Resistance; Noninsulin-dependent Diabetes Mellitus
Keywords: Cardiovascular Disease; Inflammation; Insulin Resistance; Type 2 DM
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Inflammation; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — salicylsalicylic acid; Sodium Salicylate; polynoxylin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo
- Salsalate Therapy (Active Comparator): Salsalate
  Interventions: Drug: Salsalate

INTERVENTIONS:
Drug: Salsalate — Participants were randomized to 12-week treatment with up to 4 g/day.
  Other Names: Amigesic; Anaflex; Argesic-SA; Disalcid; Marthritic; Mono-Gesic; Salflex; Salsitab
  Arms: Salsalate Therapy
Drug: Placebo — Participants were randomized to 12-week treatment matching the active salsalate arm.
  Arms: Placebo

SUMMARY:
The hypothesis is that salsalate therapy may be an effective and safe method to modulate inflammation in metabolically-critical tissues and thus reduce insulin resistance and its related complications.

The objectives of the study are to (1) determine whether salsalate therapy improves insulin resistance in subjects with IGT and changes in glucose area under the curve following a standard oral glucose tolerance test (OGTT); (2) determine whether salsalate therapy reduces a) plasma levels of a variety of well established inflammatory proteins and b) mononuclear cell inflammatory activity to provide evidence of reduced systemic and tissue inflammation, respectively; and (3)also determine whether salsalate therapy improves parameters of cardiovascular disease risk, including features of metabolic syndrome (fasting glucose, triglycerides, HDL, and blood pressure) as well as endothelial dysfunction.

DETAILED DESCRIPTION:
Recent studies demonstrate an important role for sub-acute, chronic inflammation in the development of insulin resistance, type 2 diabetes mellitus (T2 DM) and cardiovascular disease (CVD). A broad body of data indicate that obesity and high fat or "Western" diets activate sub-acute inflammatory processes in fat and liver tissue as well as in mononuclear cells. The inflammatory mediators produced by these tissues and cells promote the development of insulin resistance both locally and at distant sites such as skeletal muscle. These same inflammatory mediators may also increase the risk for CVD. Work from our labs indicate that Nuclear Factor-kappa B (NF-kB), an inflammatory master switch for a multitude of proinflammatory genes and pathways, is activated in fat and liver by obesity and high fat diets. We have also noted similar NF-kB activation in monocytes and macrophages in similar conditions of nutritional excess. It has become evident that salicylates inhibit the NF-kB regulatory protein IKKB (inhibitor of Kappa B Kinase) and we have subsequently demonstrated their ability to downregulate NF-kB activation in each of these above tissues in animals. Moreover, by inhibiting the IKKB/NF-kB pathway, salicylates appear to ameliorate insulin resistance and its associated metabolic abnormalities and potentially provide a new approach for pharmacologic treatment of T2 DM as well as individuals with conditions such as impaired glucose intolerance (IGT) to prevent their progression to diabetes. Preliminary results from a two-week trail is T2 DM patients indicated that high-dose aspirin(ASA,~7g/day) improved glucose metabolism and associated risk factors. While this was as important first step towards proof-of-principle, the risk of severe gastrointestinal bleeding associated with high-dose ASA precludes broader use. Salicylate in its prodrug form of salsalate(Disalcid), is much safer than ASA(as it does not irritate the gastric mucosa nor alter bleeding times). We have now conducted several preliminary short-term in individuals with IGT or T2 DM as well in obese insulin resistant subjects and have demonstrated that salsalate in doses of 3.5-4.5g/d provides similar blood salicylate levels as high dose ASA and induces similar clinical and metabolic benefits over the 2-4 weeks study duration. Therefore, in vitro, animal and human clinical studies all support the concept that inhibiting the IKKB/NF-kB pathway with salsalate is a feasible approach to reducing insulin resistance. This study will more fully characterize the metabolic benefits of high dose salsalate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female veterans between the age of 21-75 who have IFG (impaired fasting glucose) and/or IGT

Exclusion Criteria:

* any diabetes therapy in the prior 12-months period
* any acute illness
* Ongoing high dose aspirin or Salsalate Therapy
* history of GI bleeding
* hearing problems
* poor vascular access, prior pancreatitis, uncontrolled hypertension, pregnancy, renal disease or anemia

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reaven, MD, Principal Investigator — Carl T. Hayden VA Medical Center
Locations (1):
- Carl T. Hayden VA Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Result] Goldfine AB, Conlin PR, Halperin F, Koska J, Permana P, Schwenke D, Shoelson SE, Reaven PD. A randomised trial of salsalate for insulin resistance and cardiovascular risk factors in persons with abnormal glucose tolerance. Diabetologia. 2013 Apr;56(4):714-23. doi: 10.1007/s00125-012-2819-3. Epub 2013 Jan 31. PMID 23370525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were veterans aged 21-75 years with impaired fasting glucose (i.e. ≥5.6 but <7 mmol/l) or impaired glucose tolerance (2 h glucose values ≥7.8 but <11.1 mmol/l) during a standard 2 h 75 g OGTT. Study participants were recruited from clinics and hospitals throughout the Phoenix and Boston VA Health Care systems.
Pre-assignment Details: After enrolment there were 1 week screening, 3 week single-masked placebo run-in (to assess compliance) and 12 week randomised, double-masked treatment periods, with participants randomised 1:1 to receive salsalate or placebo. 78 individuals entered the run-in phase.
Groups:
- Salsalate: Salsalate therapy (Caraco Pharmaceutical Labs, Detroit, MI, USA) was initiated at 3.0 g/day and increased at weeks 2 and 4 of the treatment period to 3.5 and 4.0 g/day, respectively, in divided doses twice daily, as tolerated.
Period: Overall Study
Arm/Group | Placebo | Salsalate
Started | 37 | 34
Received Study Medication | 36 | 34
Completed | 30 | 29
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: Seventy-eight individuals entered the placebo run-in phase. Of these, 71 were randomised and 70 returned to receive study medication
Groups:
- Salsalate Therapy: Salsalate therapy, double-masked. Salsalate (Caraco Pharmaceutical Labs, Detroit, MI, USA) was initiated at 3.0 g/day and increased at weeks 2 and 4 of the treatment period to 3.5 and 4.0 g/day, respectively, in divided doses twice daily, as tolerated for 12 weeks total.
- Total: Total of all reporting groups
Arm/Group | Placebo | Salsalate Therapy | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 60 (6) | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 35 | 32 | 67
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 34 | 70
Insulin sensitivity [Mean (Standard Deviation); unit: mg/ kg . min] — Whole-body insulin sensitivity was estimated from glucose infusion rate (GIR) during last 30 min of euglycemic-hyperinsulinemic clamp.
  mg/ kg . min | 4.08 (1.46) | 3.8 (1.0) | 3.93 (1.27)
Oral Glucose Tolerance Test [Mean (Standard Deviation); unit: mg/dl. min] — Area Under the Curve Measurement
  mg/dl. min | 167 (21) | 165 (17) | 166 (19)
Fasting glucose [Mean (Standard Deviation); unit: mg/dl] | 105 (12) | 103 (10) | 104 (11)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systemic Glucose Disposal- Glucose Infusion Rates
Description: Participants were admitted to the Clinical Research Units at 06:00-08:00 hours after an overnight fast. Euglycaemic-hyperinsulinaemic clamps were conducted at baseline and at the end of the study. Because salsalate therapy appears to decrease insulin clearance leading to higher circulating insulin levels during the clamp, we reduced the infusion rate of insulin in the active treatment arm by 20% (from 100 to 80 mUm-2 min-1) at the study end. Insulin solutions were prepared by the site pharmacist so that study staff remained blinded to drug assignment. Whole-body insulin sensitivity was estimated from glucose infusion rate (GIR) during last 30 min of insulin infusions.
Time Frame: 3 months
Population: analysis was performed on all participants with available baseline and final clamp studies
Measure: Median (95% Confidence Interval); unit: percent change from baseline
Groups:
- Placebo: Placebo: Matching placebo
- Salsalate Therapy: Salsalate: Salsalate therapy
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 29 | 29
percent change from baseline | 1 [-39 to 56] | 6 [-20 to 61]
Statistical Analysis 1: Comparison: Placebo vs Salsalate Therapy; Paired comparisons (follow-up vs baseline) and unpaired group comparisons were performed by Student's t tests or Wilcoxon signed rank tests; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Glucose Area Under the Curve in These Subjects
Time Frame: 3 months
Population: analysis was performed on all participants with available baseline and final clamp studies
Measure: Mean (Standard Deviation); unit: mmol/l/hr
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 30 | 28
mmol/l/hr | 8.98 (1.19) | 8.74 (1.33)

3. Secondary Outcome: Plasma CRP
Description: Plasma C-reactive protein was measured by PVAHS clinical laboratory. Data are reported as change from baseline at 8 and 12 weeks.
Time Frame: 8 and 12 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: mg/l
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 36 | 34
mg/l
  Change in CRP at 8 weeks | 0 [-2.3 to 4.1] | -0.8 [-8 to 4.5]
  Change in CRP at 12 weeks | -0.1 [-2.6 to 3.6] | -.3 [-5.6 to 4.5]

4. Secondary Outcome: Endothelial Function
Description: Endothelial-mediated arterial responses using peripheral arterial tonometry (PAT; Itamar Medical, Caesarea, Israel).
Time Frame: Baseline and 12 weeks
Population: Analysis was performed on all participants with available baseline and final clamp studies
Measure: Mean (Standard Error); unit: index
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 26 | 27
index
  Pat Index baseline | 1.8 (.5) | 1.9 (.5)
  Pat Index 12 week | 1.7 (.5) | 1.7 (.6)

5. Secondary Outcome: Plasma Interleukin 6
Description: Plasma IL-6 was measured by ELISA. Data are reported as change from baseline at 8 and 12 weeks.
Time Frame: 8 and 12 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: pg/ml
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 36 | 34
pg/ml
  Change in IL-6 at 8 weeks | 0.1 [-0.5 to 0.9] | 0 [-0.2 to 0.4]
  Change in IL-6 at 12 weeks | 0.2 [-0.3 to 0.7] | 0 [-0.2 to 0.7]

6. Secondary Outcome: Plasma sVCAM
Description: Plasma soluble VCAM was measured by ELISA. Data are reported as change from baseline at 8 and 12 weeks.
Time Frame: 8 and 12 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: ng/ml
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 36 | 34
ng/ml
  Change in sVCAM at 8 weeks | -12 [-162 to 75] | -5 [-105 to 272]
  Change in sVCAM at 12 weeks | 9 [-145 to 166] | 171 [7 to 320]

7. Secondary Outcome: Plasma Adiponectin
Description: Plasma soluble Adiponectin was measured by ELISA. Data are reported as change from baseline at 8 and 12 weeks.
Time Frame: 8 and 12 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: μg/ml
Arm/Group | Placebo | Salsalate Therapy
Number analyzed (Participants) | 36 | 34
μg/ml
  Change in adiponectin at 8 weeks | -0.5 [-1.1 to 0.3] | 1.3 [-0.1 to 2.1]
  Change in adiponectin at 12 weeks | -0.1 [-1 to 1.7] | 1.2 [-0.4 to 2.8]

ADVERSE EVENTS:
Time Frame: 14 weeks (12 weeks active treatment + 2-week follow-up).
Groups:
- Placebo: Placebo: Matching placebo The frequency of tinnitus was relatively low (n=4 for salsalate, n= 2 for placebo), only one instance was graded > mild. Gastrointestinal complaints did not differ between groups (n= 8 for salsalate, n=5 for placebo). No hypoglycaemia occurred.
- Salsalate Therapy: Salsalate: Salsalate therapy The frequency of tinnitus was relatively low (n=4 for salsalate, n= 2 for placebo), only one instance was graded > mild. Gastrointestinal complaints did not differ between groups (n= 8 for salsalate, n=5 for placebo). No hypoglycaemia occurred.
Arm/Group | Placebo | Salsalate Therapy
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 7/36 | 12/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Salsalate Therapy (N=34)
tinnitus (Ear and labyrinth disorders) | 2 (2) | 4 (4) — The frequency of tinnitus was relatively low (n=4 for salsalate, n= 2 for placebo), only one instance was graded > mild
nausea (Gastrointestinal disorders) | 5 (5) | 8 (8)

LIMITATIONS AND CAVEATS:
Since we did not measure endogenous glucose production and lipolysis, the effects on hepatic glucose and lipid metabolism deserve further study. Sufficient numbers of women were not included, with which to confidently extend these results to women

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No